CLINICAL TRIAL: NCT02421705
Title: Visceral Sensitivity in IBD and IBS: Role of Inflammation, Immune Activity and Genetic Factors
Brief Title: Visceral Sensitivity in IBD (Irritable Bowel Disease) and IBS (Irritable Bowel Syndrome)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Guy Boeckxstaens, Prof. Dr., KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S51573
Record Dates: First submitted 2013-07-31; First posted 2015-04-21 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: IBS; Ulcerative Colitis, Active; Ulcerative Colitis, Remission (3a: With IBS Symptoms, 3b: Without IBS Symptoms); Healthy Controls; Crohn's Disease, Active; Crohn's Disease, Remission (6a: With IBS Symptoms, 6b: Without IBS Symptoms)
MeSH Terms: conditions — Colitis, Ulcerative; Motor Activity; Crohn Disease | interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sample collection (Other): Collection of blood, feces samples, sample of nasal mucosa and biopsies (rectum and colon descendens), questionnaires and performance of rectal sensitivity measurement (barostat), MR scan of brain and transit measurement of colon
  Interventions: Other: Sample collection

INTERVENTIONS:
Other: Sample collection — Collection of blood, feces samples, sample of nasal mucosa and biopsies (rectum and colon descendens), questionnaires and performance of rectal sensitivity measurement (barostat), MR scan of brain and transit measurement of colon

SUMMARY:
Aim:

More insight in pathogenesis of IBS and IBD. Samples are collected in context of an European research project.

DETAILED DESCRIPTION:
Methods:

Sample collection in healthy subjects, IBD and IBS patients:

* biopsy of rectum and colon descendens
* blood sample collection
* collection of sample of nasal mucosa
* feces collection
* questionnaires
* rectal barostat sensitivity measurement
* transit measurement of colon
* MR scan of brain

ELIGIBILITY:
Inclusion Criteria:

For group 1: IBS

1. Irritable Bowel Syndrome (IBS) (ROME III criteria)
2. No obvious organic explanation for the IBS symptoms
3. Medication which affects the gastrointestinal motility or perception should be stopped at least 24 hours before the study

Group 2: active ulcerative colitis 1. diagnosis of ulcerative colitis (Confirmed by at least one sigmoidoscopy) 3. Medication which affects the gastrointestinal motility or perception should be stopped at least 24 hours before the study

Group 3: ulcerative colitis in remission (3a: with IBS symptoms, 3b: without IBS symptoms)

1. diagnosis of ulcerative colitis (Confirmed by at least one sigmoidoscopy)
2. remission is confirmed by at least one sigmoidoscopy
3. Medication which affects the gastrointestinal motility or perception should be stopped at least 24 hours before the study

   Only for group 3a:
4. Rome III criteria for IBS

Group 4: Healthy controls No abdominal (pain) complaints.

Group 5: active Crohn's disease

1. diagnosis of Crohn's disease (Confirmed by at least one sigmoidoscopy) 3. Medication which affects the gastrointestinal motility or perception should be stopped at least 24 hours before the study

Group 6: Crohn's disease in remission (6a: with IBS symptoms, 6b: without IBS symptoms)

1. diagnosis of Crohn's disease (Confirmed by at least one sigmoidoscopy)
2. remission is confirmed by at least one sigmoidoscopy
3. Medication which affects the gastrointestinal motility or perception should be stopped at least 24 hours before the study

Exclusion Criteria:

For all groups:

1. co-morbidity: severe kidney- and/or liver disease or thyroid abnormalities and impaired clotting
2. Abdominal chirurgy (except for an uncomplicated appendectomy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99999999 (Estimated)
Dates: Start 2010-02; Primary Completion 2099-01 (Estimated); Study Completion 2099-01 (Estimated)

PRIMARY OUTCOMES:
differences in visceral sensitivity in different study groups (Visceral sensitivity will me measured by performing a rectal barostat test) | at time of investigation (rectal barostat test), Day 1
  Visceral sensitivity will me measured by performing a rectal barostat test

SECONDARY OUTCOMES:
immune activity (measuring release of mest cell mediators in rectal biopsies, measuring parameters of immune activity in blood) | at time of investigation (rectal biopsy), Day 1
  measuring release of mest cell mediators in rectal biopsies, measuring parameters of immune activity in blood (for example by stimulating Peripheral Blood Mononuclear Cells)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Boeckxstaens, MD, Principal Investigator — Catholic University Leuven and Universitary Hospitals Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium